CLINICAL TRIAL: NCT04326985
Title: A Randomized Control Clinical Trial to Evaluate the Efficacy of Intra-articular Injections of Mesenchymal Stem Cells Versus Hyaluronic Acid in Patients Affected by Osteoarthritis of the Knee
Brief Title: RCT Mesenchymal Stem Cells Versus Hyaluronic Acid in OA Knee):
Acronym: MSC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OA MSC Study protocol v 1.4
Record Dates: First submitted 2020-03-27; First posted 2020-03-30 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous Mesenchymal Stem Cells Treatment (MSCs) (Experimental): The MSCs treatment group patients will receive an intra-articular injection of a mesenchymal stem cell (MSCs) suspension in the affected knee.
  The treatment will be carried out after the patient has received a blood test and clinically evaluated at T0.
  T0: Beginning of the study, blood test and bone marrow aspiration. T30: Intra-articular injection of MSCs T44: Adverse events follow up 2 weeks after intra-articular injection (by phone)
  Interventions: Biological: Autologous Mesenchymal Stem Cells Treatment (MSCs)
- Hyaluronic acid (HA) (Active Comparator): The patient will be given a single intra-articular injection of hyaluronic acid sodium salt, Synvisc-One (TRB Chemedica Ltd.) The hyaluronic acid will be purchased for the patient from the manufacturer or from the pharmacy of the hospital.The intra-articular injection will be carried out after the patient has received a clinical evaluation at T0.
  T0: Beginning of the study T30: Intra-articular injection of Synvisc-One (HA) T44: Adverse events follow up 2 weeks after intra-articular injection (by phone)
  Interventions: Drug: Hyaluronic acid (HA)

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells Treatment (MSCs) — The MSCs treatment group patients will receive an intra-articular injection of a mesenchymal stem cell (MSCs) suspension in the affected knee.
  Arms: Autologous Mesenchymal Stem Cells Treatment (MSCs)
Drug: Hyaluronic acid (HA) — The HA group patient will be given a single intra-articular injection of hyaluronic acid sodium salt, Synvisc-One (TRB Chemedica Ltd.)
  Arms: Hyaluronic acid (HA)

SUMMARY:
The purpose of this study is to evaluate the therapeutic effect of adult autologous mesenchymal stem cells (abbreviated as MSCs) in patients with osteoarthritic knee and compare to intra articular injection of Synvisc-One.

DETAILED DESCRIPTION:
Study Participants:

This study will involve patients affected by osteoarthritis who comply with the inclusion and exclusion criteria. 30 patients, between the age of 18 and <65, will be enrolled in the study and randomized into three groups to receive either an injection of MSCs, hyaluronic acid (HA) or no injection.

Type of Study: This is a randomized control study.

Treatment method: Each patient will randomly be assigned to one of the following treatment groups:

Group A) Mesenchymal stem cells (MSCs) Group B) Hyaluronic acid (HA) Group C) No injection

Treatment:

Group A) Autologous Mesenchymal Stem Cells Treatment (MSCs) The MSCs treatment group patients will receive an intra-articular injection of a mesenchymal stem cell (MSCs) suspension in the affected knee.

The treatment will be carried out after the patient has received a blood test and clinically evaluated at T0.

T0: Beginning of the study, blood test and bone marrow aspiration. T30: Intra-articular injection of MSCs T44: Adverse events follow up 2 weeks after intra-articular injection (by phone)

Group B) Hyaluronic acid (HA) The patient will be given a single intra-articular injection of hyaluronic acid sodium salt, Synvisc-One (TRB Chemedica Ltd.) The hyaluronic acid will be purchased for the patient from the manufacturer or from the pharmacy of the hospital.

The intra-articular injection will be carried out after the patient has received a clinical evaluation at T0.

T0: Beginning of the study T30: Intra-articular injection of Synvisc-One (HA) T44: Adverse events follow up 2 weeks after intra-articular injection (by phone)

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and < 65
* Radiological evidence of osteoarthritis with Kellgren and Lawrence grade 2 and 3
* Patients on a pain level equal to or higher than 5 on a VAS scale of 10

Exclusion Criteria:

* Previous cases of alcoholism or drug abuse
* Pregnancy and breast-feeding
* Serious pathologies such as carcinoma or autoimmune disease
* Hypersensitivity toward Hyaluorinc Acid
* Undergoing steroid-based systemic therapy or interrupted since less than 1 month
* Significant hematologic diseases
* Mechanical instability, ligamentous laxity/deficiency or gross deformity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | One year
  Clinical Questionnaire Assessment Tool. Score 80-100 = Excellent, Score 70-79 = Good, Score 60-69 = Fair, Score below 60 = Poor
Knee Society Function Score | One year
  Clinical Questionnaire Assessment Tool. Score from 100 to -20. The higher the score, the better the knee function outcome.
Magnetic resonance image (MRI) and X-ray assessment | One year
  Radiological assessment of the knee joint

SECONDARY OUTCOMES:
Health related quality of life score (HRQoL) - SF36 | One year
  Questionnaire Assessment
Western Ontario and McMaster Osteoarthritis Index (WOMAC) | One year
  Questionnaire Assessment
Visual Analogic Scale (VAS) pain evaluation | One year
  Questionnaire Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided